CLINICAL TRIAL: NCT04781920
Title: Follow-up of Anterior Cruciate Ligament Reconstruction
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN162021/CHUSTE
Record Dates: First submitted 2021-02-25; First posted 2021-03-04 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Anterior Cruciate Ligament; reconstruction; Operative report; Consultation report; Isokinetic tests; Clinical surveys
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients having undergone an Anterior Cruciate Ligament (ACL) reconstruction: Patients having undergone an ACL reconstruction will be included.
  Interventions: Other: datas collection

INTERVENTIONS:
Other: datas collection — data collection in history medical : operative report, clinical examination, questionnaires, imaging, isokinetic tests

SUMMARY:
Rupture of Anterior Cruciate Ligament (ACL) is a common pathology, but is subject to variability of associated lesions, surgical management and rehabilitation.

DETAILED DESCRIPTION:
In this study, a collect data of patients having undergone an Anterior Cruciate Ligament (ACL) reconstruction in order to evaluate the clinical, functional and morphological results of this intervention, in order to improve the management of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients having undergone an Anterior Cruciate Ligament (ACL) reconstruction

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having undergone an Anterior Cruciate Ligament (ACL) reconstruction will be included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Analysis of Magnetic Resonance Imaging (MRI) results | Pre-operative and Month: 12
  Collected in medical records

SECONDARY OUTCOMES:
Analysis of operative report results | Month: 12
  Collected in medical records
Analysis of consultation report | pre-operative and Months: 1,5 , 3, 6, 12
  Collected in medical records
Analysis of isokinetic tests | Months: 9, 12
  Collected in medical records
Analysis of clinical surveys | pre-operative and Months: 3, 6, 12
  Collected in medical records

CONTACTS AND LOCATIONS:
Overall Officials: Thomas NERI, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No